CLINICAL TRIAL: NCT00762398
Title: Evaluation of the Accuracy and Precision of the Masimo Labs Pulse-Hemoglobin-Meter Monitor in Surgical Patients
Status: Terminated | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Masimo Labs (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-6221
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Adult Patient Undergoing Major Surgery
Keywords: Major surgery, excpected blood loss, arterial line

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for the measurement of Hct, and ABG
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult patient undergoing a surgery: Adult patient undergoing a surgery in the supine position and require an arterial line for anesthesia/surgery purposes
  Interventions: Device: Masimo hemoglobin-meter; Biological: drawing blood sample

INTERVENTIONS:
Device: Masimo hemoglobin-meter — Placing a probe on the finger
Biological: drawing blood sample — drawing a blood sample less that 0.5 mL each time, for around 10-12 times along the surgery (depends on surgical time)

SUMMARY:
The Masimo monitor can measure hemoglobin level noninvasively and accuratly

DETAILED DESCRIPTION:
Blood hemoglobin concentration is a very common and essential test to assess patient well being and the need for blood transfusion. In the perioperative period this measurement is further more critical mainly due to the acute nature of blood loss and the need for an immediate response. Currently, hemoglobin concentration is determined by analyzing a blood sample. It requires venipuncture or arterial puncture (via an arterial line). Besides the patient discomfort there are additional disadvantages such as infection, dealing with blood product, delay with diagnosis, low update rate and cost. Masimo Labs is in the process of developing a noninvasive monitor to detect hemoglobin concentrations in real time. The monitor uses a probe placed on the patient finger that gives hemoglobin concentration continuously and noninvasively. Masimo Labs is using a technology that resembles the well accepted and clinically proven pulse-oxymeter.

The study will include surgical patients at the UCI Medical Center, preferably in cases that are known to involve major blood loss. For these cases, the anesthesia team places an arterial line for anesthesia purposes. The arterial line is used for continuous blood pressure measurements and blood draw for the assessment of several indices. We plan to compare the hemoglobin concentrations measured from blood samples to the Masimo Labs pulse-hemoglobin level readings.

ELIGIBILITY:
Inclusion Criteria:

* Adult having surgery with arterial line

Exclusion Criteria:

* Upper extremities surgery
* Pregnant women
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in UCI Medical Center undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
corrlation of up to +/-0.1 gr% of the blood analysis to the monitor reading | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Rosenbaum, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Univeristy of California Irvine Medical Center, Orange, California, United States